CLINICAL TRIAL: NCT02070627
Title: Near Infrared Fluorescence Cholangiography (NIRF-C) During Cholecystectomy Sub-Study
Brief Title: Near Infrared Fluorescence Cholangiography (NIRF-C) During Cholecystectomy -- Use in Acute Cholecystitis Sub-Study
Acronym: NIRF-C Acute
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Principal Investigator, Narula, Vimal K, MD, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011H0239S
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Acute Cholecystitis; Acute Cholangitis
Keywords: acute cholecystitis; acute cholangitis; cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIRF-C and IOC (Experimental): Each enrolled subject will undergo injection with indocyanine green (ICG), intraoperative near infrared fluorescence cholangiography (NIRF-C) and standard of care intraoperative cholangiography.
  Interventions: Drug: Indocyanine Green (ICG); Device: Near Infrared Fluorescence Cholangiography (NIRF-C)

INTERVENTIONS:
Drug: Indocyanine Green (ICG) — 60-30 minutes prior to cholecystectomy, 2.5 mg of indocyanine green (ICG) will be injected intravenously. An additional 2.5 mg of ICG may be injected intraoperatively if the fluorescence fades prior to imaging.
Device: Near Infrared Fluorescence Cholangiography (NIRF-C) — Near infrared fluorescence cholangiography will be performed intraoperatively in order to image anatomy.
  Other Names: Stryker 1488 Camera System; Stryker L9000 Light Source; Stryker 1488 Coupler; Stryker 10mm Ideal Eyes Laparoscope (0 and 30 degree)

SUMMARY:
The purpose of this study is to evaluate an imaging system using Indocyanine Green (ICG) to assist in real-time identification of anatomy during cholecystectomy (gallbladder removal) in patients with acute cholecystitis and cholangitis. We propose to define the effectiveness of NIRF-C in identifying the cystic duct junction during cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Planned laparoscopic cholecystectomy

Exclusion Criteria:

* Inability to provide informed consent
* Pregnant
* Allergy to ICG, iodine, and/or shellfish
* Lactating

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Adverse events related to use of indocyanine green (ICG) | Injection to 2 wk follow-up
  Adverse events related to the use of ICG from the time of injection through the initial post-operative clinic visit will be recorded and assessed.
Anatomic identification with NIRF-C and IOC | Intraoperative
  Anatomic identification with near-infrared fluorescence cholangiography and standard of care intraoperative cholangiography (IOC) will be used to calculate a 95% confidence interval for the effectiveness of this modality.
Procedure time | Intraoperative
  The time it takes to perform near infrared fluorescence cholangiography and standard of care intraoperative cholangiography will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Vimal K Narula, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States